CLINICAL TRIAL: NCT02614976
Title: Incidences of Cuff-related Trauma After Noninvasive Blood Pressure Measurement Between With and Without Padding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Mingkwan Wongyingsinn, MD, Dr., Siriraj Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SIRB157
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No padding before application of blood pressure cuff
- Padding (Experimental): Padding before application of blood pressure cuff
  Interventions: Device: Padding

INTERVENTIONS:
Device: Padding — Padding webrill (Covidian) TM 6"
  Arms: Padding

SUMMARY:
Padding with cuff during blood pressure is expected to reduce number of skin crease or petechiae incidence.

DETAILED DESCRIPTION:
Objective Primary Outcome : incidences of skin crease or petichiae after noninvasive blood pressure measurement ievery 5 minutes for 1 hour Secondary Outcome : factor related truma after noninvasive blood pressure measurement.

ELIGIBILITY:
Inclusion Criteria:

* Health volunteer age > 18 or patients

Exclusion Criteria:

* Peripheral vascular disease
* Difference of blood pressure both arms > 15 mmHg
* Acute dermal cappillary rupture
* Phlebitis
* Skin necrosis
* Acute radial nerve injury
* Deep vein thrombosis
* Rumpel-Leede phenomenon
* Compartment syndrome

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Complication of a non-invasive blood pressure cuff | 5 minutes after completion of non-invasive blood pressure measuring
  Petechiae and skin crease

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, M.D., Study Director — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkoknoi, Bangkok, Thailand